CLINICAL TRIAL: NCT00664768
Title: A Prospective, Randomized, DB Controlled Study to Evaluate the Nutritional Safety (Growth) of an Amino Acid Based Formula With Prebiotics and Probiotics in Infants Diagnosed With Cow Milk Allergy, With or Without Other Food Allergies.
Brief Title: A Growth and Hypoallergenicity Study of a New Formula for Infants With Cow Milk Allergy
Acronym: CMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia North America (Industry)
Collaborators: Nutricia Liverpool (Industry); Danone Institute International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT0131
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Cow Milk Allergy
Keywords: hypoallergenicity; Cow Milk Allergy; DBPCFC; Stool microflora; Stool characteristics
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- New Neocate (Experimental): new Neocate
  Interventions: Dietary Supplement: new Neocate
- Neocate Infant (Active Comparator): Neocate Infant formula
  Interventions: Dietary Supplement: Neocate Infant

INTERVENTIONS:
Dietary Supplement: Neocate Infant — minimum of 8 fl. oz daily
  Arms: Neocate Infant
Dietary Supplement: new Neocate — minimum of 8 fl oz daily
  Arms: New Neocate

SUMMARY:
This study involves the use of 2 different Neocate formulas: a control formula called Neocate Infant and a test Neocate formula. These kinds of formulas are for use in children from birth to 8 months of age with Cow Milk Allergy (CMA), other food allergies, and other gastrointestinal disorders. The purpose of this study is to compare the control and test Neocate formulas for safety, tolerability, and effectiveness (in promoting growth) when used in subjects with CMA.

This study will also look at the test Neocate formula to see if it is hypoallergenic when used in subjects with CMA.

DETAILED DESCRIPTION:
Infants who qualify will begin a 7-day milk protein elimination diet that excludes all milk or products which contain milk. Parents will be asked to keep a food diary of everything the child eats during the week following the Screening Visit. During this week, the child can continue to drink their current hypoallergenic formula.

Subjects will be assessed at seven study visits at baseline, two weeks, four weeks and then monthly until the end of the study period, where the following will be assessed:

Study Visit 1 (Day -7): Baseline

This will be carried out at entry to the trial to collect baseline data; at this visit subjects will under go the following assessments:

Assess Patient suitability Obtain Informed Consent Obtain Subject number Perform physical exam and clinical assessment Medical history and assessment including SCORing Atopic Dermatitis assessment (SCORAD) Obtain weight, length and head circumference Collect a 9ml venous blood sample The following is to analysed by the central lab; Plasma total protein/albumin and prealbumin Blood urea nitrogen, electrolytes and creatinine Complete blood count with differential Alkaline phosphatase. Serum Iron, Total Iron Binding Capacity and Ferritin Plasma fatty acid analysis Provide stool lab kits and explain to parent/caregiver how to collect stool sample during the pre-evaluation week Provide one-week subject diary (Subject Diary 1) and instruct parent/caregiver on how to complete record, clinical symptoms and stool characteristics (frequency, consistency and color) in subject diary.

Provide the one-week Food Frequency Diary A and instruct the parent/caregiver on how to complete this assessment Provide information on following a milk protein exclusion diet, with or without the exclusion of other allergenic food proteins as advised by the subject's physician Record all concomitant medications taken within two weeks prior to the Baseline Visit

Study Visit 2 (Day 0): Once subjects have completed the pre-evaluation period subjects will undergo the following assessment:

Review Subject Diary 1 and Food Frequency Diary A, for study compliance Randomisation assignment to one of the two study formulas Perform physical exam and clinical assessment Obtain weight, length/height and head circumference Provide two-week subject diary (Subject Diary 2a) and instruct parent/caregiver on how to record clinical symptoms and stool characteristics in subject diary.

Provide the one-week Food Frequency Diary B and instruct the parent/caregiver on how to complete this assessment Collect stool sample that was obtained in previous week at home

Phone review (Day 7)

Subjects will be reviewed at this time point by telephone to review if any clinical symptoms have occurred while ingesting study formula. If it is determined by the Principal Investigator that the subject has had any clinically significant reaction(s) to the study formula, the subject must return to the clinic for evaluation. Subjects will progress to Phase II and continue feeding with the formula they have consumed as part of the seven-day, post-challenge feeding period.

Study Visit 3 (Day 14): Two weeks on formula

Once subjects have been consuming their assigned formula for a two week period the following assessment will be carried out:

Obtain weight, length and head circumference Collect Subject Diary 2a and Food Frequency Diary B Review of open feeding period and presence of any clinical symptoms Provide one-week subject diary (Subject Diary 3) to be completed the week before returning for Visit 4 and instruct parent/caregiver on how to record, clinical symptoms and stool characteristics in subject diary.

Provide three-day Food Diary 1 to be completed the week before returning for visit 4 and instruct parent/caregiver on how to complete the food records Instruct parent to collect stool sample during the week before study Visit 4. Review study product requirement and dispense as necessary

Study Visit 4 (Day 28): One month on formula

Once subject have been consuming test formula for one month they will undergo the following assessment:

Perform clinical assessment and SCORAD Obtain weight, length and head circumference Obtain stool sample collected by parent Collect and review Subject Diary 3 and Food Diary 1 Review study product requirement and dispense as necessary

Study Visit 5 (Day 56): Two months on formula Obtain weight, length and head circumference Provide 3 day subject diary (Subject Diary 4) to be completed in the following week and instruct parent/caregiver on how to record clinical symptoms and stool characteristics in subject diary Provide three-day Food Diary 2 to be completed in the following week and instruct parent/caregiver on how to complete the food records Review study product requirement and dispense as necessary

Study Visit 6 (Day 84): Three months on formula Obtain weight, length and head circumference Collect Subject Diary 4 and Food Diary 2 Provide one week subject diary (Subject Diary 5) to be completed in the week prior to the final study visit and instruct parent/caregiver on how to complete the food records, clinical symptoms and stool characteristics in subject diary Provide three-day Food Diary 3 to be completed in the week prior to the final study visit and instruct parent/caregiver on how to complete the food records Instruct parent to take stool sample during the week before the final study visit Review study product requirement and dispense as necessary

Study Visit 7 (Day 112): Final visit - four months on formula or Early Termination Perform clinical assessment and SCORAD Obtain weight, length and head circumference Obtain stool sample collected by parent Collect and review Subject Diary 5 and Food Diary 3 Collect blood sample Ensure Parents/caregivers have returned all diaries to the appropriate clinician at each center Study personnel will review the forms with the parents/caregivers Parents/caregivers will return all partial and unopened cans of the test formula

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged from birth to 8 months old with documented allergy to cow milk protein are eligible to enter the study. Subjects with other IgE or non IgE mediated allergies to food in addition to milk protein (e.g. multiple food allergy or an eosinophilic disorder) are also eligible to enter the study. However all subjects must have a confirmed allergy to milk confirmed by one of the following criteria, within two months prior to the baseline visit:

   * Positive double-blind placebo controlled food challenge with cow milk
   * A confirmed history of acute severe reaction after isolated accidental ingestion with a positive test result for IgE antibody
   * Confirmed history of a reaction to cow milk protein with CM-specific IgE of >15kU/L for children over two years and > 5kU/L for children under two years.
   * Confirmed clinical history of a reaction to cow milk protein with a positive skin prick test with a resulting wheal diameter greater or equal to 3mm.
   * No confirmed clinical history of a reaction to cow milk protein subjects with a positive skin prick test with a resulting wheal diameter greater or equal to 8mm for children over 2 years and greater or equal to 6mm for children under 2 years.
   * For children with an Allergic Eosinophilic Gastroenteritis (AEG), documentation of eosinophilic infiltration and resolution of symptoms on a diet that restricted cow milk (and other foods) with reoccurrence after re-administration of cow milk.
2. Written informed consent / ability to give informed consent.
3. These subjects are expected to consume a minimum intake of test formula to ensure an average daily intake, which provides at least 50% of their daily energy requirements,

Exclusion Criteria:

All subjects

1. Infants <5lb 8oz at birth
2. Infants < 37 weeks gestation
3. Infants with severe concurrent illness or major congenital malformations
4. Suspected or documented systemic or congenital infections (e.g. human immunodeficiency virus)
5. Unable to adhere to protocol instructions due to non compliance of parent or caregiver
6. Investigator's uncertainty about the willingness or ability of the patient to comply with the protocol requirements
7. Participation in any other studies involving investigational products concomitantly or within twenty eight days prior to entry into the study
8. An infant of any personnel connected with the study
9. Infants whose parent/caregiver is younger than the legal age of consent
10. For these subjects the dietary consumption of other sources of prebiotics or probiotics is prohibited two weeks prior to inclusion in the study and during the study period.
11. These subjects must not have received systemic antibiotics in the previous two weeks prior to entry into the study.

Ages: 1 Day to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2008-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is attained growth (i.e. incremental gains in weight) over the study period. | 4 months
  The primary endpoint is attained growth (i.e. incremental gains in weight) over the study period. Length and head circumference measures will also be collected and analysed. Both the growth velocities of the group as a whole (cross-sectional group data) and individuals (longitudinal individual data) will be reviewed and analysed. In assessing group data, comparisons of increments per unit of time will be made. Due to the varying ages of the subjects recruited to the study, growth measures will be concerted to z-scores using an appropriate reference population to allow a meaningful comparison of the ability of the formulas to promote growth. In assessing the growth of individual infants, data will be plotted on National Centre for Health Statistics (NCHS) growth charts and assessed qualitatively.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Mourmans, Study Director — Study Mgr Nutricia Research - Centre for Specialised Nutrition
Locations (22):
- United States (22):
  - Pendleton Pediatrics, Chandler, Arizona
  - Visions Clinical Research - Tucson, Tucson, Arizona
  - Children's Investigational Research Program, LLC (CHIRP), Bentonville, Arkansas
  - Children's Hospital, LA, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Rosario B. Retino, MD, Inc, Ontario, California
  - Choc Psf, Amc, Orange, California
  - Nemours Children's Clinic, Jacksonville, Florida
  - Alzein Pediatrics, Evergreen Park, Illinois
  - Regional Research Specialists, LLC, Shreveport, Louisiana
  - Craig A. Spiegel, M.D., Bridgeton, Missouri
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Weill Cornell Medical College, New York, New York
  - Asheboro Research Associates, Asheboro, North Carolina
  - Duke University, Durham, North Carolina
  - Pediatrics, PLLC, Holly Springs, North Carolina
  - John Panuto, M.D., Middleburg Heights, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - PI-Coor Clinical Research, LLC, Burke, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Advanced Pediatrics, Vienna, Virginia

REFERENCES:
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765
- [Derived] Harvey BM, Eussen SRBM, van Helvoort A, Harthoorn LF. Cow's Milk Allergic Infants on Elemental Formula Maintain Adequate Mineral Status Despite Using Acid-suppressive Drugs. J Pediatr Gastroenterol Nutr. 2019 Nov;69(5):e147-e148. doi: 10.1097/MPG.0000000000002469. No abstract available. PMID 31425366
- [Derived] Burks AW, Harthoorn LF, Van Ampting MT, Oude Nijhuis MM, Langford JE, Wopereis H, Goldberg SB, Ong PY, Essink BJ, Scott RB, Harvey BM. Synbiotics-supplemented amino acid-based formula supports adequate growth in cow's milk allergic infants. Pediatr Allergy Immunol. 2015 Jun;26(4):316-22. doi: 10.1111/pai.12390. PMID 25845680